CLINICAL TRIAL: NCT00084799
Title: A Multiple-Dose Targeting Study of hu3S193 in Patients With Small Cell Lung Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Progressive Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-015; MSKCC 04-012 (Other: MSKCC); CDR0000365621 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer (SCLC)
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- hu3S193 10 mg/m2 (Experimental): Patients with small cell lung cancer tumors confirmed to have Lewis Y expression were enrolled to receive 4 weekly injections of hu3S193 at a dose of 10 mg/m2. The dose of hu3S193 given on Weeks 1 and 4 was trace-labeled with 6-8 millicurie (mCi) of indium-111 (111In).
  Interventions: Biological: monoclonal antibody hu3S193
- hu3S193 20 mg/m2 (Experimental): Patients with small cell lung cancer tumors confirmed to have Lewis Y expression were enrolled to receive 4 weekly injections of hu3S193 at a dose of 20 mg/m2. The dose of hu3S193 given on Weeks 1 and 4 was trace-labeled with 6-8 millicurie (mCi) of indium-111 (111In).
  Interventions: Biological: monoclonal antibody hu3S193

INTERVENTIONS:
Biological: monoclonal antibody hu3S193

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: This phase I trial is studying the side effects of monoclonal antibody therapy in treating patients with progressive small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the targeting, tissue distribution, and pharmacokinetics of monoclonal antibody hu3S193 in patients with progressive small cell lung cancer (SCLC).

Secondary

* Determine the immunogenicity of of monoclonal antibody hu3S193 in patients with progressive small cell lung cancer (SCLC).
* Determine tumor response of monoclonal antibody hu3S193 in patients with progressive small cell lung cancer (SCLC).
* Determine the safety of tof monoclonal antibody hu3S193 in patients with progressive small cell lung cancer (SCLC).

OUTLINE: This is an open-label, pilot study.

Patients received monoclonal antibody hu3S193 (mAb hu3S193) intravenously (IV) over 30 minutes on day 1 of weeks 1-4. Patients also received indium-111 (111In) radiolabeled hu3S193 IV over 30 minutes on day 1 of weeks 1 and 4 and then underwent gamma camera imaging. Treatment continued in the absence of disease progression or unacceptable toxicity.

Patients were followed at 1 and 4 weeks, every 3 months for 1 year, and then every 6-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

Small cell lung cancer, pathologically confirmed. Measurable disease, including at least one lesion measuring ≥ 2 cm that has not been previously irradiated.

Progression of disease after one, two, or three prior chemotherapy regimens. At least 4 weeks since the last chemotherapy or radiation treatment. Karnofsky performance status ≥ 70% (ECOG 0 or 1).

The following laboratory results within the last 2 weeks prior to study day 1:

White Blood Cell Count (WBC) ≥ 3,500/mm3; Platelet count ≥ 100 x 10^9/L; Serum creatinine ≤ 2.0 mg/dL; Serum bilirubin ≤ 2.0 mg/dL; International normalized ratio (INR) ≤ 1.3; Women of childbearing potential with confirmed negative quantitative serum HCG on the day of administration of study agent.

Negative stool guaiac test (read by laboratory). Tumor tissue positive for Lewis Y expression.

Exclusion Criteria:

Clinically significant cardiac disease (New York Heart Association Class III/IV).

Uncontrolled brain or leptomeningeal metastases. GI bleed within the preceding 6 months. Patients with history of receiving mouse monoclonal antibody. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.

Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-07-26 (Actual); Primary Completion 2006-01-25 (Actual); Study Completion 2006-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Chaitanya R. Divgi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Krug LM, Milton DT, Jungbluth AA, Chen LC, Quaia E, Pandit-Taskar N, Nagel A, Jones J, Kris MG, Finn R, Smith-Jones P, Scott AM, Old L, Divgi C. Targeting Lewis Y (Le(y)) in small cell lung cancer with a humanized monoclonal antibody, hu3S193: a pilot trial testing two dose levels. J Thorac Oncol. 2007 Oct;2(10):947-52. doi: 10.1097/JTO.0b013e3181560dcc. PMID 17909358

RESULTS

PARTICIPANT FLOW:
Groups:
- hu3S193 10 mg/m2: Patients with small cell lung cancer tumors confirmed to have Lewis Y expression were enrolled to receive 4 weekly injections of hu3S193 at a dose of 10 mg/m2. The dose of hu3S193 given on Weeks 1 and 4 was trace-labeled with 6-8 mCi of indium-111 (111In).
- hu3S193 20 mg/m2: Patients with small cell lung cancer tumors confirmed to have Lewis Y expression were enrolled to receive 4 weekly injections of hu3S193 at a dose of 20 mg/m2. The dose of hu3S193 given on Weeks 1 and 4 was trace-labeled with 6-8 mCi of indium-111 (111In).
Period: Overall Study
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of hu3S193.
Groups:
- Total: Total of all reporting groups
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Confirmation of Tumor Targeting as Measured by the Number of Patients With Assessable Lesions Greater Than or Equal to 2 cm Measured by FDG-PET and SPECT Imaging.
Description: Gamma camera imaging, including planar scans and single-photon emission computed tomography (SPECT) scans, were carried out immediately following completion of infusion and on two subsequent occasions during the next 6 days after the infusions of 111In-hu3S193 on weeks 1 and 4. A pretreatment FDG-positron emission tomography PET/CT scan was performed within 2 weeks of study entry per standard clinical methods for comparison with gamma camera imaging. FDG-PET/ CT scans and 111In planar and SPECT scans were evaluated for extent of disease and antibody targeting, respectively. Lesions on FDG-PET/CT scans were considered positive if uptake of radiotracer was visually greater than surrounding tissue, with a standard uptake value greater than 3.
Time Frame: 28 days
Population: Patients who received at least one dose of hu3S193.
Measure: Count of Participants; unit: Participants
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

2. Secondary Outcome: Mean Half-life (T1/2) as Measured by 111In-hu3S193 Radioactivity
Description: Blood samples for analysis of radioactivity and serum concentration of hu3S193 were obtained immediately before and 5, 60, and 120 minutes post-infusion, before and after imaging on day 2, and on days 3 and 5 after completion of the 111In-hu3S193 infusion in weeks 1 and 4. Pharmacokinetics was calculated using WinNonLin (Pharsight Co., Mountain View, CA). A two-compartment model was fitted to individually labeled infusions for each patient using unweighted nonlinear least squares to calculate pharmacokinetic parameters.
Time Frame: 4 weeks (days 1, 2, 3, and 5; weeks 1 and 4)
Population: Patients who received at least one dose of hu3S193.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
hours
  T½α | 13.28 (11.02) | 7.45 (7.06)
  T½β | 126.22 (35.35) | 129.60 (51.93)

3. Secondary Outcome: Mean Volume of Distribution of Central Compartment (V1) as Measured by 111In-hu3S193 Radioactivity
Description: as for outcome 2
Time Frame: 4 weeks (days 1, 2, 3, and 5; weeks 1 and 4)
Population: Patients who received at least one dose of hu3S193.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
mL | 3040.78 (565.38) | 3468.07 (686.79)

4. Secondary Outcome: Mean Clearance (CL) as Measured by 111In-hu3S193 Radioactivity
Description: as for outcome 2
Time Frame: 4 weeks (days 1, 2, 3, and 5; weeks 1 and 4)
Population: Patients who received at least one dose of hu3S193.
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
mL/hour | 28.83 (15.32) | 30.81 (10.18)

5. Secondary Outcome: Mean Area Under the Curve (AUC) as Measured by 111In-hu3S193 Radioactivity
Description: as for outcome 2
Time Frame: 4 weeks (days 1, 2, 3, and 5; weeks 1 and 4)
Population: Patients who received at least one dose of hu3S193.
Measure: Mean (Standard Deviation); unit: hours*g/mL
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
hours*g/mL | 859.97 (347.19) | 1327.00 (465.47)

6. Secondary Outcome: Immunogenicity of hu3S193 as Measured by the Number of Patients With Human Anti-human Antibodies (HAHA) After Treatment With hu3S193.
Description: Blood samples to measure human anti-human antibody (HAHA) assessments were obtained at baseline and each week before hu3S193 dosing. Measurement of immune responses to hu3S193 in patient blood samples was analyzed using a BIACORE (Piscataway, NJ) instrument using surface plasmon resonance (SPR).
Time Frame: 4 weeks (pre-dose, weeks 1, 2, 3, and 4)
Population: Patients who received at least one dose of hu3S193.
Measure: Count of Participants; unit: Participants
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
Participants
  Number of Patients with HAHA | 0 | 0
  Number of Patients without HAHA | 5 | 5

7. Secondary Outcome: Number of Patients With Tumor Responses After Treatment With hu3S193 as Measured by RECIST
Description: Tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria (Therasse P et al. 2000).
Time Frame: up to 28 days
Population: Patients who received at least one dose of hu3S193.
Measure: Count of Participants; unit: Participants
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
Number analyzed (Participants) | 5 | 5
Participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 0 | 0
  PD | 5 | 5

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: All adverse events (AEs) occurring during the study were to be documented in the source records and on the respective AE Case Report Form (CRF). Adverse events which occurred prior to the first administration of study drug were documented on the Pre-existing symptoms CRF page, thereafter, they were documented on the Adverse Event CRF page. Adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 3.0, published April 16, 2003).
Arm/Group | hu3S193 10 mg/m2 | hu3S193 20 mg/m2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hu3S193 10 mg/m2 (N=5) | hu3S193 20 mg/m2 (N=5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hu3S193 10 mg/m2 (N=5) | hu3S193 20 mg/m2 (N=5)
Blood creatinine (Investigations) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Hemoglobin (Investigations) | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
International normalised ratio (Investigations) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Activated partial thromboplastin time (Investigations) | 1 | 0
Alanine aminotransferase (Investigations) | 2 | 2
Aspartate aminotransferase (Investigations) | 2 | 2
Blood alkaline phosphatase (Investigations) | 1 | 2
Blood creatine phosphokinase (Investigations) | 1 | 0
Chest pain (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Hyperbillirubinemia (Hepatobiliary disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Platelet count (Investigations) | 1 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
White blood cell count (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No